CLINICAL TRIAL: NCT03604913
Title: Aortic Valve-sparing Root Replacement Operation Versus Bentall Operation - Early and Midterm Outcomes
Brief Title: Aortic Valve Sparing Root Replacement Versus Bentall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Kamel Abd-Elnaim Hussein, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Valve sparing versus Bentall
Record Dates: First submitted 2018-07-12; First posted 2018-07-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Aortic Root Aneurysm; Aortic Root Dissection
Keywords: Valve sparing aortic root replacement
MeSH Terms: conditions — Aortic Root Aneurysm; Dissection, Ascending Aorta

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A(aortic valve sparing operation) (Active Comparator): Undergo aortic valve sparing root replacement operation
  Interventions: Procedure: Aortic valve sparing operation
- B(Bentall operation) (Active Comparator): Undergo Bentall operation
  Interventions: Procedure: Bentall operation

INTERVENTIONS:
Procedure: Aortic valve sparing operation — Aortic valve sparing instead of replacement during aortic root replacement
  Arms: A(aortic valve sparing operation)
Procedure: Bentall operation — Aortic root replacement with replacement of aortic valve
  Arms: B(Bentall operation)

SUMMARY:
This study was designed to evaluate the hypothesis that the operative and midterm results of valve-sparing aortic root replacement are equivalent to those of the Bentall.

Objective 1:

Evaluate short-term (one-to-six months) and mid-term (six-to-forty-eight months) results of aortic valve-sparing procedures.

Objective 2:

Compare the results of aortic valve-sparing procedures with the group of patients undergoing Bentall procedures during the same period.

Objective 3:

Assess outcomes of both procedures through evaluation of postoperative:

A) primary outcome measures:

1. Intraoperative or intrahospital death.
2. Reexploration for bleeding.
3. Reoperation rate.
4. Grade of aortic valve regurgitation (0-4).

B)secondary outcome measures:

1. Grade of aortic valve regurgitation (0-4).
2. Mean gradient on the aortic valve(mmHg).
3. Thromboembolism / bleeding.
4. Prosthetic/native valve endocarditis.
5. 2-year mortality

DETAILED DESCRIPTION:
The aortic root is a complex structure whose single components are of paramount importance in assuring proper functioning of the aortic valve. In fact, opening and closing behaviors of the aortic leaflets are regulated by the interaction of the various components of the aortic root as well as by the characteristics of blood flow.

Operation was the only possible surgical solution for diseases involving the sinuses of Valsalva and the aortic valve. Even in experienced hands, the perioperative mortality was not insignificant. However, since the introduction of the exclusion technique, the mortality and major morbidity of aortic root replacement have seen a dramatic decline. In recent years, groups focused on aortic disease have reported elective operative mortality less than 5%, with a marked decline in the incidence of stroke, hemorrhage, and other major postoperative complications.

The composite graft replacement, as originally reported by Bentall and De Bono in 1968, has become a milestone in proximal aortic surgery, by providing the solution to a surgical problem that was a formidable challenge for that era. From the original report, many relevant scientific papers continued to address both the disease (dilatation or dissection of the proximal aorta, involving the aortic root and, often, the aortic valve) and its surgical correction. This ongoing attention led to several major refinements of the original technique and to the development of improved prosthetic material. All these efforts were aimed at the solution of two major problems affecting the original inclusion-wrapping technique: pseudoaneurysm formation (usually at the site of coronary anastomosis) and transprosthetic bleeding due to excessive porosity of the vascular prosthesis. For many years, however, little attention was paid to the fact that, in many instances, the aortic valve was intrinsically healthy, and nonetheless was substituted, thus unnecessarily exposing the patient to the risk of valve-related complications.

The analysis of the normal anatomy and physiology of aortic root is the basis for establishing the surgical transition, in selected cases, from aortic root replacement to aortic valve-sparing operation. In 1983, however, Dr Yacoub addressed the issue of aortic insufficiency secondary to dilatation of the sinotubular junction and he proposed to resect the entire diseased aortic wall, preserving the valve with its commissural posts. A properly tailored vascular prosthesis, with three semicircular tongues, was then sutured to a small rim of the aortic wall just above the aortic annulus, following its three-cusp, crown-shaped line. The entire aortic root was therefore remodelled, thus justifying the appellation of remodelling technique, with reconstruction of a bulged root and a well defined sinotubular junction. Approximately 10 years later, Dr David introduced the aortic valve-sparing reimplantation technique by means of which the valve remnants prepared in a similar manner were reimplanted inside a cylindrical Dacron conduit.

The introduction of techniques for valve-sparing aortic root replacement over 20 years ago has allowed for the preservation of healthy aortic valve in patients with severely diseased aortic roots. Moreover, an attempt is made to reconstruct as closely as possible all anatomic components of the aortic root, thus restoring the physiologic behaviour of the aortic valve leaflets within the reshaped root. By maintaining native aortic valve function, potential adverse events related to the use of either a mechanical or a bioprosthetic valve are avoided, including eliminating the lifelong burden of anticoagulation or the risk of structural valve deterioration.

As such, valve-sparing aortic root replacement is an attractive therapy for aortic root pathology with preservation of the native aortic valve. Limited data exist comparing valve-sparing aortic root replacement and conventional aortic root replacement with a composite valve-conduit. Furthermore, these studies are limited by small patient numbers, selection bias.

ELIGIBILITY:
Inclusion Criteria:

1. Ascending aorta or aortic root aneurysm(size more than 5 cm or 4.5 cm in Marfan syndrome).
2. Ascending aorta or aortic root dissection.
3. With or without aortic regurgitation
4. Good condition of aortic cusps.

Exclusion Criteria:

1. The left ventricular ejection fraction less than 40 %.
2. Previous aortic valve replacement.
3. Aortic stenosis.
4. Patients with extensive aortic root destruction because of aortic root infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects who die | 30 days
  Number of subjects who die either intraoperative or intrahospital

SECONDARY OUTCOMES:
Grade of aortic valve regurgitation | 1,6 months and 1,2 years
  Grade of postoperative aortic valve regurgitation by echocardiography
Mean gradient(mmgh) on the aortic valve | 1,2 years
  Mean gradient(mmgh) on the aortic valve by echocardiography
Thromboembolism/bleeding | 6 months and 1,2 years
  Number of subjects who present by Thromboembolism/bleeding
Prosthetic/native valve endocarditis | 6 months and 1,2 years
  Number of subjects who present with prosthetic/native valve endocarditis

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Nady, Lecturer, Study Chair — Assist university
Locations (1):
- Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Majumder PP, St Jean PL, Ferrell RE, Webster MW, Steed DL. On the inheritance of abdominal aortic aneurysm. Am J Hum Genet. 1991 Jan;48(1):164-70. PMID 1985458
- [Background] Gillum RF. Epidemiology of aortic aneurysm in the United States. J Clin Epidemiol. 1995 Nov;48(11):1289-98. doi: 10.1016/0895-4356(95)00045-3. PMID 7490591
- [Background] De Paulis R, Bassano C, Bertoldo F, Chiariello L. Aortic valve-sparing operations and aortic root replacement. J Cardiovasc Med (Hagerstown). 2007 Feb;8(2):97-101. doi: 10.2459/01.JCM.0000260209.73097.f4. PMID 17299290
- [Background] Bentall H, De Bono A. A technique for complete replacement of the ascending aorta. Thorax. 1968 Jul;23(4):338-9. doi: 10.1136/thx.23.4.338. PMID 5664694
- [Background] Zehr KJ, Orszulak TA, Mullany CJ, Matloobi A, Daly RC, Dearani JA, Sundt TM 3rd, Puga FJ, Danielson GK, Schaff HV. Surgery for aneurysms of the aortic root: a 30-year experience. Circulation. 2004 Sep 14;110(11):1364-71. doi: 10.1161/01.CIR.0000141593.05085.87. Epub 2004 Aug 16. PMID 15313937
- [Background] Mataraci I, Polat A, Kiran B, Caliskan A, Tuncer A, Erentug V, Kirali K, Isik O, Yakut C. Long-term results of aortic root replacement: 15 years' experience. Ann Thorac Surg. 2009 Jun;87(6):1783-8. doi: 10.1016/j.athoracsur.2009.03.046. PMID 19463595
- [Background] Etz CD, Bischoff MS, Bodian C, Roder F, Brenner R, Griepp RB, Di Luozzo G. The Bentall procedure: is it the gold standard? A series of 597 consecutive cases. J Thorac Cardiovasc Surg. 2010 Dec;140(6 Suppl):S64-70; discussion S86-91. doi: 10.1016/j.jtcvs.2010.07.033. PMID 21092800
- [Background] Kouchoukos NT, Wareing TH, Murphy SF, Perrillo JB. Sixteen-year experience with aortic root replacement. Results of 172 operations. Ann Surg. 1991 Sep;214(3):308-18; discussion 318-20. doi: 10.1097/00000658-199109000-00013. PMID 1834031
- [Background] Sarsam MA, Yacoub M. Remodeling of the aortic valve anulus. J Thorac Cardiovasc Surg. 1993 Mar;105(3):435-8. PMID 8445922
- [Background] David TE, Feindel CM. An aortic valve-sparing operation for patients with aortic incompetence and aneurysm of the ascending aorta. J Thorac Cardiovasc Surg. 1992 Apr;103(4):617-21; discussion 622. PMID 1532219
- [Background] Gaudino M, Lau C, Munjal M, Avgerinos D, Girardi LN. Contemporary outcomes of surgery for aortic root aneurysms: A propensity-matched comparison of valve-sparing and composite valve graft replacement. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1120-9.e1. doi: 10.1016/j.jtcvs.2015.07.015. Epub 2015 Jul 10. PMID 26234456
- [Background] Coselli JS, Volguina IV, LeMaire SA, Sundt TM, Connolly HM, Stephens EH, Schaff HV, Milewicz DM, Vricella LA, Dietz HC, Minard CG, Miller DC; Aortic Valve Operative Outcomes in Marfan Patients Study Group. Early and 1-year outcomes of aortic root surgery in patients with Marfan syndrome: a prospective, multicenter, comparative study. J Thorac Cardiovasc Surg. 2014 Jun;147(6):1758-66, 1767.e1-4. doi: 10.1016/j.jtcvs.2014.02.021. Epub 2014 Feb 8. PMID 24655904
- [Background] Toeg H, Chan V, Rao RV, Chan KL, Ruel M, Mesana T, Boodhwani M. Contemporary midterm echocardiographic outcomes of Bentall procedure and aortic valve sparing root replacement. Ann Thorac Surg. 2014 Aug;98(2):590-6. doi: 10.1016/j.athoracsur.2014.04.121. Epub 2014 Jun 24. PMID 24968770
- [Background] Tourmousoglou C, Rokkas C. Is aortic valve-sparing operation or replacement with a composite graft the best option for aortic root and ascending aortic aneurysm? Interact Cardiovasc Thorac Surg. 2009 Jan;8(1):134-47. doi: 10.1510/icvts.2008.186544. Epub 2008 Oct 21. PMID 18940830
- [Background] Lim JY, Kim JB, Jung SH, Choo SJ, Chung CH, Lee JW. Surgical Management of Aortic Root Dilatation with Advanced Aortic Regurgitation: Bentall Operation versus Valve-sparing Procedure. Korean J Thorac Cardiovasc Surg. 2012 Jun;45(3):141-7. doi: 10.5090/kjtcs.2012.45.3.141. Epub 2012 Jun 7. PMID 22708080